CLINICAL TRIAL: NCT05086549
Title: A Multicenter, Prospective, Observational Study to Evaluate the Renoprotective Effect of Fimasartan in Patients With Diabetic Kidney Disease and Proteinuria
Brief Title: An Observation Study to Evaluate the Renoprotective Effect of Fimasartan in Patients With DKD and Proteinuria
Acronym: FINALE
Status: Completed | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BR-FMS-OS-407
Record Dates: First submitted 2021-09-23; First posted 2021-10-21 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Diabetic Kidney Disease; Proteinuria; Hypertension,Essential
Keywords: Fimasartan; Proteinuria
MeSH Terms: conditions — Diabetic Nephropathies; Proteinuria; Essential Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to observe changes in various indicators of renal function, such as proteinuria at different time points: short-term (Week 8), 6 months (Week 26), and a year (Week 52), in patients with DKD and hypertension, who are given antihypertensives containing fimasartan, in an actual clinical environment where a variety of patient characteristics are reflected.

DETAILED DESCRIPTION:
This prospective observational study is conducted in about 5 medical institutions located in Korea, which are equal to or larger than a hospital, and patients with type 2 diabetic kidney disease (proteinuria with an ACR of 10 mg/g or higher), who are being administered or plan to be administered with antihypertensives containing fimasartan for essential hypertension, are enrolled as the subjects. Each of the subjects shall undergo follow-up for about a year (52 weeks). After explaining the purpose, method, scope of information to be collected, and procedure of this study to potential subjects, the investigator shall obtain the written consent for voluntary participation and set the day when the antihypertensive containing fimasartan is administered as the baseline. If the fimasartan-based antihypertensive treatment is already ongoing, only the patients within 6 weeks from the baseline shall be considered as the subjects. In this case, data from between the baseline and the time of the written consent shall be collected retrospectively. This study is an observational study, and the drugs which are administered during the study period and the medical procedures shall be in accordance with the clinical judgment of the investigator. It is a rule that no unnecessary intervention shall be imposed on the subjects by this study protocol.

The scope of data to be collected during this study period is as follows.

* Demographic information
* Disease information (diabetes, hypertension, renal disease, other past medical history and intercurrent diseases)
* Physical measurements (height and weight)
* Clinic blood pressure measurements
* Laboratory test results
* Antihypertensives, hypoglycemic agents, and other concomitant drugs
* Fimasartan-related adverse drug reactions and serious adverse drug reactions
* Death information (if applicable)

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged 19 or older
* Those who were diagnosed with type 2 diabetes and have been being given stable doses of hypoglycemic agents for 8 weeks or longer
* Those in whom albuminuria was found to meet one of the following criteria two times before the administration of the antihypertensive treatment containing fimasartan (results (baseline values) within 4 weeks before the administration of antihypertensives must be ACR or AER results)

  * An albumin/creatinine ratio (ACR) of 10 mg/g or higher or
  * An albumin excretion rate (AER) of 10 mg/day or higher or
  * A proteinuria/creatinine ratio (PCR) of 70 mg/g or higher or
  * A urine dipstick result of trace to 1+ or higher
* Those who plan to be given antihypertensive treatment containing fimasartan for essential hypertension or are being given the treatment (in this case, those with an administration period of 6 weeks or lower can be enrolled)
* Those with records of clinical systolic blood pressure of 140 mmHg or higher or diastolic blood pressure of 85 mmHg or higher before the antihypertensive treatment containing fimasartan or at the time of the treatment. The following additional criteria shall be applied depending on age and the presence of comorbidities.

  * Aged younger than 65: Systolic blood pressure of 130 mmHg or higher or diastolic blood pressure of 80 mmHg or higher shall be applied to those with cardiovascular disease or an ACR or AER of 30 mg/g or higher.
  * Aged 65 or older: Regardless of comorbidities, systolic blood pressure of 140 mmHg or higher or diastolic blood pressure of 90 mmHg or higher shall be applied.
* Patients who agreed in writing to the Personal Information Collection and Usage Agreement after listening to the explanation of the objective, method, etc. of this observational study

Exclusion Criteria:

* Patients who are suspected of or confirmed with secondary hypertension
* Those diagnosed with type 1 diabetes or secondary diabetes
* Patients undergoing kidney dialysis or patients who received kidney transplants or those for whom kidney dialysis or kidney transplants are planned
* If angiotensin converting enzyme inhibitors (ACEI) or renin inhibitors are used in conjunction or are planned to be used in conjunction
* Patients with moderate to severe hepatic dysfunction (ALT and/or AST of over three times the upper limit of normal) or patients with biliary tract obstruction
* Pregnant and breast-feeding women
* Those who were administered with drugs for clinical studies within 12 weeks from the enrollment or those who plan on participating in other clinical studies while participating in this study
* Other subjects who are considered inappropriate to participate in the study by the investigator's decision

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetic kidney disease and proteinuria (urine ACR of 10 mg/g or higher)
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
Rate of change in albuminuria (urine ACR) | Week 8
  The descriptive statistics (number of subjects, average, standard deviation, median, minimum value, quartile, and maximum value) regarding the rate of change in albuminuria (urine ACR) at the baseline, on Week 8, and on Week 8 compared to the baseline shall be obtained

SECONDARY OUTCOMES:
Quantity of change in albuminuria (urine ACR) | Week 8
  The descriptive statistics (number of subjects, average, standard deviation, median, minimum value, quartile, and maximum value) regarding the quantity of change in albuminuria (urine ACR) at the baseline, on Week 8, and on Week 8 compared to the baseline shall be obtained
Rate of change in albuminuria (urine ACR) | Week 26, Week 52
  The descriptive statistics (number of subjects, average, standard deviation, median, minimum value, quartile, and maximum value) regarding the rate of change in albuminuria (urine ACR) at each time point, on Week 26 and Week 52 compared to the baseline shall be obtained
Rate of change in proteinuria (urine PCR) | Week 8, Week 26, Week 52
  The descriptive statistics (number of subjects, average, standard deviation, median, minimum value, quartile, and maximum value) regarding the rate of change in proteinuria (urine PCR) at each time point, on Week 8, Week 26, and Week 52 compared to the baseline shall be obtained

CONTACTS AND LOCATIONS:
Overall Officials: MyungSook Hong, Study Director — Boryung Pharmaceutical Co., Ltd
Locations (1):
- Severance hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No